CLINICAL TRIAL: NCT02325258
Title: Assessment of a Proposed Microbiological Alert and Its Impact on a Sepsis Campaign
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emilio Bouza (Other)
Responsible Party: Sponsor-Investigator, Emilio Bouza, Head of Department, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MICRO.HGUGM.2012-001
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Sepsis
Keywords: Sepsis diagnosis; Sepsis drug therapy; Sepsis outcome
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone call (Experimental): Telephone call to physicians in charge of patients who have just had blood cultures drawn. Diagnostic and therapeutic recommendations to physicians in charge.
  Interventions: Other: Telephone call
- No telephone call (No Intervention): control arm: no intervention

INTERVENTIONS:
Other: Telephone call — Aug-Dec 2012. Prospective study in patients who had blood cultures drawn and sent to the Microbiology Lab during the morning shift (9 am to 3 pm, Mon- Fri) to evaluate sepsis recognition. The investigators allocated 300 patients to 2 groups of 150 patients each, by opportunity sampling: patients whose clinical history number ended in odd numbers were assigned to group A (intervention) and those whose clinical history number ended in even numbers were assigned to group B (no intervention, control group). For patients in group A, the investigators attempted a telephone contact with the physician and/or nurse in charge and an interview, issuing recommendations regarding the convenience of further biochemical, microbiological or extra radiologic tests, and management and antimicrobial therapy.
  Arms: Telephone call

SUMMARY:
The aim of the present study was to evaluate the ability of health-care professionals in addressing sepsis, and the impact of a telephone call upon receival of blood cultures in the clinical microbiology department, from a clinical microbiologist, in the early management of sepsis.

DETAILED DESCRIPTION:
Sepsis is one of the major challenges of modern medicine. It is an important health problem with a high incidence, morbidity and mortality that affects population worldwide. Without an early recognition and a prompt management, patients can develop more severe stages of the disease and even death. An appropriate and aggressive management can significantly improve outcomes. Thus, it is necessary to develop early warning systems of sepsis in the hospital.

In recent years, several campaigns and guidelines have been developed to help health care professionals in the management of sepsis. However, these have mainly focused on management protocols for severe sepsis and septic shock in intensive care units or emergency departments. To the best of the investigators knowledge, none of these have examined in depth either the impact of a sepsis alert system in general wards, nor the impact of a telephone call from a specialist in Clinical Microbiology, upon blood culture request, in the early recognition of sepsis.

The aim of the present study was to evaluate the ability of health-care professionals in addressing sepsis, and the impact of a telephone call upon receival of blood cultures in the clinical microbiology department, from a clinical microbiologist, in the early management of sepsis.

For this, the investigators performed a prospective study based on telephone calls followed by a phone interview to physicians and nurses in charge of patients whose blood cultures had just been received at the clinical microbiology department in a tertiary hospital.

ELIGIBILITY:
In-patients with blood cultures drawn and sent to the Microbiology laboratory, regardless of patient allocation (eg., emergency department, intensive care units, general wards)

Opportunity sampling: patients whose clinical history number ended in odd numbers were assigned to group A (intervention) and patients whose clinical history number ended in even numbers were assigned to group B (no intervention, control group).

Inclusion Criteria:

* Patients who had blood cultures drawn and sent to the Microbiology Laboratory, during the morning shift (from 9 am to 3 pm, Monday to Friday)
* Patients >/=18 years old

Exclusion Criteria:

* Patients <18 years old
* Patients with a recent bacteremic episode with no subsequent negative blood cultures
* In-patients with blood cultures drawn to whom the telephone call had already been performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Sepsis recognition in patients who had blood cultures drawn | 72 h
  Use of diagnostic resources and antimicrobial consumption

SECONDARY OUTCOMES:
Health care professionals who correctly identify a case of sepsis | 72 h

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Bouza Santiago, MD, PhD, Principal Investigator — Servicio de Microbiología y Enfermedades Infecciosas; Eleonora Bunsow, MD, PhD, Study Director — Servicio de Microbiología y Enfermedades Infecciosas; Marcela González Del Vecchio, MD, Study Chair — Servicio de Microbiología y Enfermedades Infecciosas; Carlos Sánchez, PharmD, Study Chair — Servicio de Microbiología y Enfermedades Infecciosas; Patricia Muñoz García, MD, PhD, Study Chair — Servicio de Microbiología y Enfermedades Infecciosas; Almudena Burillo, MD, PhD, Study Chair — Servicio de Microbiología y Enfermedades Infecciosas
Locations (1):
- Servicio de Microbiologia y Enfermedades Infecciosas, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Bunsow E, Vecchio MG, Sanchez C, Munoz P, Burillo A, Bouza E. Improved Sepsis Alert With a Telephone Call From the Clinical Microbiology Laboratory: A Clinical Trial. Medicine (Baltimore). 2015 Sep;94(39):e1454. doi: 10.1097/MD.0000000000001454. PMID 26426609